CLINICAL TRIAL: NCT04110821
Title: Quality of Life After Conservative and Surgical Treatment of Pelvic Organ
Brief Title: Quality of Life After Conservative and Surgical Treatment of Pelvic Organ Prolapse
Acronym: LOLIPOP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-01190
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Pelvic Organ Prolapse; Quality of Life; Incontinence
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study that gives baseline and follow-up information, that does not directly influence the allocation of patients to various treatment Options (conservative and surgical therapy of Pelvic Organ Prolapse) but the knowledge gained of the data will help to develop treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

- Pelvic Organ Prolapse (POP)

Exclusion Criteria:

* < 18 years
* Patients unable to understand an informed consent
* Patients unwilling to participate
* emergency operations
* pregnancy
* Overactive Bladder without descensus
* Stool incontinence without POP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study all patients with POP being treated at the study site are subject to inclusion. This concerns patients with different symptoms of POP such as urine or fecal incontinence, chronic obstipation, dysfunction of the bowel evacuation, micturition disorder, chronic pelvic pain, complaints associated to pelvic floor descent and pelvic organ prolapse. They also may have combinations of these symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2019-09-15 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
symptom change assessed by German Pelvic Floor Questionnaire (GPFQ) | before therapy and up to 5 years post-therapy
  Change in the symptom scores assessed by the German Pelvic Floor Questionnaire (GPFQ) by at least 1.0 points 6 months post-therapy.
  The GPFQ does contain the domains bladder function, bowel function, prolapse and sexual symptoms. In each domain a total of 10 points may be reached. The maximum symptom score for the entire questionnaire are 40 points. The minimal symptom score is 0 points. The minimal important difference (MID) for patients with Pelvic Organ Prolapse (POP) is 1.0 points. A decrease of the symptom score by at least 1 point reflects a meaningful improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Steinemann, PD Dr. med., Principal Investigator — University Hospital Basel, Clarunis
Locations (1):
- University Hospital Basel/Dep. of Visceral Surgery (Clarunis), Basel, Switzerland